CLINICAL TRIAL: NCT01057290
Title: Stat3 Activation as a Potential Prognostic Marker and Therapeutic Target in Pediatric AML
Brief Title: Studying Biomarkers in Cell Samples From Young Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AAML10B16; COG-AAML10B16 (Other: Children's Oncology Group); CDR0000664194 (Other: Clinical Trials.gov); NCI-2011-02206 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: childhood acute myeloid leukemia/other myeloid malignancies
MeSH Terms: conditions — Leukemia | interventions — Gene Expression Profiling; Flow Cytometry; Immunologic Techniques

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — cell samples
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis
Genetic: protein expression analysis
Other: fluorescence activated cell sorting
Other: immunologic technique
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how well patients will respond to treatment.

PURPOSE: This research study is looking at biomarkers in cell samples from young patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To characterize Stat3 signaling pathway activity in primary tissue samples from pediatric patients with acute myeloid leukemia to determine the percentage of samples with increased activity and to better understand the mechanisms leading to increased activity.
* To evaluate the presence of constitutive Stat3 activation and the sensitivity of Stat3 activation to low and high doses of cytokines.
* To evaluate the expression levels of Stat3 protein as well as upstream and downstream regulators of Stat3 activation.
* To classify tissue samples according to a Stat3-activation pattern, and to correlate this result with event-free survival and overall survival in order to determine whether increased Stat3 phosphorylation at diagnosis predicts poor outcome.

OUTLINE: Cryopreserved cell samples are collected for laboratory analysis, including immunoblotting, fluorescence activated cell sorting (FACS), and protein analysis.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of pediatric acute myeloid leukemia

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosis of pediatric acute myeloid leukemia
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Correlation of the Stat3 response category (constitutive, low-dose responsive, high-dose responsive, or unresponsive) with clinical data, including event-free and overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Michele S. Redell, MD, PhD, Principal Investigator — Texas Children's Cancer Center